CLINICAL TRIAL: NCT03277157
Title: The Effects of Bifidobacterium Animalis Ssp. Lactis B94 on Gastrointestinal Function in Adults With Prader-Willi Syndrome: A Randomized, Double-blind Study
Brief Title: B. Lactis B94 Effects of Gastrointestinal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB201701976
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Quality of Life

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The B. lactis and placebo will be provided in identical capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Bifidobacterium animalis ssp. lactis B94 at 15 billion CFUs per capsule
  Interventions: Dietary Supplement: B. lactis B94
- Placebo (Placebo Comparator): Placebo veggie capsule.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. lactis B94 — A probiotic dose of 15 billion per capsule.
  Other Names: Bifidobacterium animalis ssp lactis B94
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo capsule
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the effect of daily consumption of Bifidobacterium animalis ssp lactis B94 (B. lactis B94) on stool frequency, gastrointestinal (GI) transit time, and gastrointestinal symptoms in adults with Prader-Willi syndrome. Participants (18-75 years old, n=36) will be recruited and enrolled in a 20-week randomized, placebo-controlled, crossover study. Study participants will be randomized to B. lactis B94 or placebo each for a 4-week period, preceded by a 4-week baseline and followed by 4-week washouts. Participants will complete daily questionnaires about stool frequency and stool form (transit). Dietary intake will also be assessed. A total of 5 stools (one in each period) will be collected for exploratory microbiota analysis. It is hypothesized that the B. lactis B94 will increase stool frequency, decrease the percentage of slow transit stools, and improve GI symptoms

DETAILED DESCRIPTION:
Probiotics have been shown to improve symptoms of constipation by decreasing gastrointestinal transit time, increasing stool frequency, and normalizing stool form. A 20-week randomized, double-blinded, placebo-controlled crossover study will be carried out. Participants will complete a 4-week baseline period during which stool frequency, stool consistency (transit time), and gastrointestinal symptoms will be collected by paper questionnaire, and participants will collect a single stool. Dietary intake data (3-day) will be obtained during the baseline period. Participants will be randomized on or about day 29 and will consume Bifidobacterium animalis ssp lactis B94 (B. lactis B94) or placebo for 4 weeks, followed by a 4-week washout, 4 weeks on the alternative, and second 4-week washout. Participants will be randomized by sealed envelope method, prepared by a UF faculty member not affiliated with the study.

During the intervention and washout periods, participants will complete daily questionnaires to assess stool frequency and form (Bristol Stool Form Scale). Furthermore, they will complete Gastrointestinal Symptom Rating Scale (GSRS) at weeks 4, 8, 12, 16 and 20(± 3 days). During these same weeks (± 3 days) dietary intake data (28-day record) and stools will be collected (1 per period). Participants' height and weight will be taken at baseline, and weight during weeks 4, 8, 12, 16 and 20.

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to provide informed consent.
* Have confirmed diagnosis of PWS
* Are willing to have height and weight measured and provide demographic information (e.g. age, race, sex)
* Are 18-75 years of age
* Are willing to consume B. lactis B94 and placebo each for 4-week periods
* Are willing to complete a daily questionnaire throughout the 20-week period.
* Are willing to complete the Gastrointestinal Symptom Rating Scale (GSRS) monthly throughout the 20-week study
* Are willing to provide information about their dietary intake for 3-days every 4 weeks
* Are willing to provide a valid social security for study payment purposes

Exclusion Criteria:

* Have a milk protein allergy
* Are currently taking medications for diarrhea
* Are currently taking probiotics supplements and do not want to discontinue prior to the start of the baseline period (i.e. those that discontinue will be included)
* Have previously or are currently being treated for any gastrointestinal diseases such as (gastric ulcers, Crohn's, Celiac, ulcerative colitis, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 4 weeks
  Weekly stool frequency - difference between treatments

SECONDARY OUTCOMES:
Stool frequency percentage change | 4 weeks
  Weekly stool frequency: percentage change from baseline
Bristol Stool Form | 4 weeks
  Percentage slow transit (Bristol Stool Form Scale 1 and 2)
Gastrointestinal symptoms | 4 weeks
  Decrease in syndromes of Gastrointestinal Symptom Rating Scale (GSRS)
Compliance | 4 weeks
  >80% of supplement intake

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - ARC of Alachua County, Gainesville, Florida
  - UF Health Pediatrics - Gerold L. Schiebler CMS Center, Gainesville, Florida
  - Food Science and Human Nutrition Department, University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alyousif Z, Miller JL, Sandoval MY, MacPherson CW, Nagulesapillai V, Dahl WJ. The effects of Bifidobacterium animalis ssp. lactis B94 on gastrointestinal wellness in adults with Prader-Willi syndrome: study protocol for a randomized controlled trial. Trials. 2018 Apr 27;19(1):256. doi: 10.1186/s13063-018-2648-x. PMID 29703235